CLINICAL TRIAL: NCT06777251
Title: Changing the Future of Intestinal Failure in Intestinal Chronic Inflammation: Towards Innovative Predictive Factors and Therapeutic Targets.
Brief Title: Changing the Future of Intestinal Failure in Intestinal Chronic Inflammation (INT-FAIL)
Acronym: INT-FAIL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Papa Alfredo, MD, Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 5483
Record Dates: First submitted 2023-03-14; First posted 2025-01-15 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Intestinal Failure; Inflammatory Bowel Diseases; Crohn Disease
MeSH Terms: conditions — Intestinal Failure; Inflammatory Bowel Diseases; Crohn Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Investigation of predictive factors in patients with intestinal failure in crohn disease (Other): * Typing of gut microbiota, metabolome and immunological signatures (IL 1b family and GLP-2 as starting point) in patients with CD and SBS/IF and in two cohorts of patients with CD, respectively at low and high risk of SBS /IF.
  * Combining data from gut microbiota, metabolome and immunological analysis using tools based on Artificial Intelligence (AI) and Machine Learning (ML) technologies.
  * Creation of a stool Biobank of categories of patients with Crohn's disease at high risk of SBS/IF and of patients with SBS with or without clinical symptoms of IF.
  Interventions: Other: analysis of predictive factors of IF in patients with Crohn's disease through the characterization of "multiomics" parameters

INTERVENTIONS:
Other: analysis of predictive factors of IF in patients with Crohn's disease through the characterization of "multiomics" parameters — The study includes an initial evaluation in which faecal samples will be collected, a blood sample will be taken and an ileocolonoscopy with biopsies will be performed (additional biopsy in conjunction with a biopsy from clinical practice for study-specific analyses).
  Patients will then be reevaluated nine months after the initial evaluation. In particular, fecal, blood and additional biopsy samples will be collected in conjunction with clinical practice biopsy and all treatment modifications will be recorded.

SUMMARY:
This is an interventional, prospective, no profit study that will be performed at CEMAD, from FONDAZIONE POLICLINICO GEMELLI IRCCS, Rome (UO1) and U.O.C. Internal Medicine and Gastroenterology from Ospedale Brotzu di Cagliari (UO4). Adult patients with Crohn Disease (CD) and chronic intestinal insufficiency (CF) and adult patients with CD at high and low risk of CF.

DETAILED DESCRIPTION:
The study involves an initial evaluation in which faecal samples will be collected, a blood sample will be taken and an ileocolonoscopy with biopsy (additional biopsy collection at the same time as clinical practice biopsy for study-specific analysis) will be performed.

Patients will then be re-evaluated nine months after the initial evaluation. In particular, faecal, blood and additional biopsy samples will be collected at the same time as the clinical practice biopsy and any changes in treatment will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years-old and ≤ 75 years old
* Capable of expressing informed consent;
* An established diagnosis of Crohn's disease;
* Antibiotics treatment free for at least 15 days.

Exclusion Criteria:

* Age < 18 years-old and > 75 years old;
* Not capable of expressing informed consent;
* Pregnant or breastfeeding patients;
* Comorbidities including: cancer pathology present or under active treatment; coagulopathies; chronic hepatopathy, heart failure, renal failure, respiratory failure.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Estimated)
Dates: Start 2024-02-29 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-05-18 (Estimated)

PRIMARY OUTCOMES:
Predictive Factors for FH in Crohn's Disease Using Gut Microbiota Composition | 24 month
  This section focuses on characterizing the gut microbiota composition in patients with Crohn's disease at risk of SBS/IF. Advanced sequencing technologies and bioinformatics tools will be used to analyze the relative abundance of microbial species associated with SBS/IF risks.
  Unit of Measure: percentage or relative abundance of microbial taxa. Objective: To identify microbiota profiles predictive of dysbiosis and their association with SBS/IF risk factors.
Predictive Factors for FH in Crohn's Disease Using Metabolome Analysis | 24 month
  This section emphasizes the analysis of metabolic profiles. Key metabolites associated with SBS/IF risk will be quantified using mass spectrometry and other advanced chemical analysis techniques.
  Unit of Measure: metabolite concentration (e.g., µM, mM). Objective: To understand how metabolic variations influence the development of SBS/IF and support the design of targeted nutritional interventions.
Predictive Factors for FH in Crohn's Disease Using Immunological Signature Characterization | 24 month
  This section investigates the characterization of immunological biomarkers. Specific levels of the IL-1β family and GLP-2 will be measured as indicators of immune response and intestinal repair mechanisms.
  Unit of Measure: concentration (pg/mL). Objective: To identify immunological signatures associated with an increased risk of SBS/IF and optimize biomarker-based therapeutic strategies.

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Papa, MD, Principal Investigator — Fondazione Policlinico A. Gemelli IRCCS, Rome
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, Italy